CLINICAL TRIAL: NCT06458790
Title: African American Resilient Caregivers
Brief Title: Black Resilient Caregivers
Acronym: AARC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pro00111805_1
Record Dates: First submitted 2024-06-06; First posted 2024-06-14 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2024-09

CONDITIONS: Obesity, Childhood
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AARC Intervention (Experimental): This intervention will adapt an already-existing evidence-based Centering Parenting program. Investigators will not provide clinical care to participants. Investigators will also address topics that are specific to African American families. Investigators will conduct 7 90 min sessions via zoom and in person.
  Interventions: Behavioral: AARC

INTERVENTIONS:
Behavioral: AARC — This intervention will adapt an already-existing evidence-based Centering Parenting program addressing topics that are specific to African American families. There will be 7 90 min sessions via zoom. Group education topics include (parenting goals, infant feeding and sleep, self-care). Participants will complete surveys and interviews at various times to evaluate the program. The survey topics will include: parent stress, parent confidence and thoughts about the intervention. Surveys will be completed independently by participants online via redcap at a time that is convenient to them; if requested, the coordinator may complete the survey with the participant directly by phone /zoom. Interviews will be completed with a coordinator via zoom/phone.

SUMMARY:
To determine the feasibility of an intervention to promote the physical and socioemotional health of African American (AA) families.

DETAILED DESCRIPTION:
AA parents face unique racialized stressors which negatively impact their health and the health of their children. This heavy burden of chronic stress contributes to a high prevalence of anxiety and depression in AA parents. Parent stress negatively impacts child development and family health behaviors including diet and physical activity. A culturally-tailored intervention that addresses both AA parent stress and early childhood health and development has the potential to be more effective in promoting healthy family behaviors and AA parent mental health than traditional early childhood preventive care. Guided by AA parents and community members, the investigators propose to systematically co-develop a novel intervention using two frameworks: Centering and Superwoman Schema. The novel intervention will include group parent support, training in stress management and links to relevant community resources. The investigators will then determine the feasibility, acceptability, and limited efficacy of the adapted intervention in a pilot study.

ELIGIBILITY:
Inclusion Criteria:

* Identify as African American/Black
* Expecting a child due September, October or November 2024
* Feel comfortable discussing personal experiences and asking questions in front of a group of peers
* Access to zoom, preferably with video
* Live in North Carolina
* Infant and mom home within 96 hours of birth

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2024-09-20 (Actual); Primary Completion 2025-11-25 (Actual); Study Completion 2025-11-25 (Actual)

PRIMARY OUTCOMES:
Acceptability as measured by the Acceptability of Intervention Measure | 7 months
  Acceptability of Intervention Measure (modified) uses the following scale: Completely disagree / Disagree / Neither agree nor disagree / Agree / Completely agree.
  The more participants agree or completely agree, the better the outcome.
Feasibility as measured by the Acceptability of Intervention Measure | 7 months
  Acceptability of Intervention Measure - Feasibility (modified) uses the following scale: Completely disagree / Disagree / Neither agree nor disagree / Agree / Completely agree.
  The more participants agree or completely agree, the better the outcome
Semi-structured Interview | 7 months
  Semi-structured interview is measured by Qualitative Interview Questions that assess practicality, acceptability and appropriateness.

SECONDARY OUTCOMES:
Parenting Confidence | 3 months and 6 months
  Measured via Karitane Parenting Confidence Scale. Each item on the Karitane Parenting Confidence Scale is scored 0, 1, 2, or 3. There are no reverse-scored items and items have a common scoring order. That is, for each item the first response is scored 0, the second 1, and so on. Items marked not applicable are scored 2. Scores are then summed to give a total score (range = 0-45). The higher the range the better the outcome.
Parent stress | At baseline and 5 months
  Measured via perceived stress scale.
  Perceived Stress Scale score by following these directions:
  First, reverse the scores for questions 4, 5, 7, and 8. On these 4 questions, change the scores like• this: 0 = 4, 1 = 3, 2 = 2, 3 = 1, 4 = 0. Now add up the scores for each item to get a total. Individual scores on the Perceived Stress Scale can range from 0 to 40 with higher scores indicating higher perceived stress.
  * Scores ranging from 0-13 would be considered low stress.
  * Scores ranging from 14-26 would be considered moderate stress.
  * Scores ranging from 27-40 would be considered high perceived stress.
Family Empowerment | 3 months and 6 months
  Measured via the Family Empowerment Scale
  This measures scores for the subscales are simple means. Calculate the mean for each subscale by adding the scores for the subscale items that have NOT been answered "Not Applicable," and dividing by the number of questions that were answered "Never…Very Often" (1 through 5). If there are missing items (up to 3) in responses 1-5, add the scores for the subscale items, and divide by the number of answered questions.
  Add responses to all of the subscales for an overall score but be aware that each of the subscales addresses quite a different topic (Family, Service System, Community). Many published articles have employed the method of adding all items for an overall score.
  Examining each subscale score in relation to other variables of interest is another approach that may yield more specific information.
GISCOMBE SUPERWOMAN SCHEMA (SWS) QUESTIONNAIRE | At baseline and 5 months
  Measured via average scores for each SWS subscale.
  RESPONSE VALUE This is NOT TRUE for me 0 This is TRUE for me RARELY 1 This is TRUE for me SOMETIMES 2 This is TRUE for me ALL THE TIME 3
  If SWS subscale items are summed to create one SWS total, these categories can be used:
  0-35: Low SWS 36-70: Moderate SWS 71-105: High SWS
  Subscales:
  Strength (6 items):
  0-6 Low 7-12 Moderate 13-18 High
  Suppress (7 items):
  0-7 Low 8-14 Moderate 15-21 High
  Resistance (7 items):
  0-7 Low 8-14 Moderate 15-21 High
  Motivation (6 items):
  0-6 Low 7-12 Moderate 13-18 High
  Help (9 items):
  0-9 Low 10-18 Moderate 19-27 High
  SWS appraisal items should be averaged.
  RESPONSE VALUE This bothers me NOT AT ALL 0 This bothers me SOMEWHAT 1 This bothers me VERY MUCH 2
Session Evaluation | 1-7months
  Session Evaluation(modified) uses the following scale: Strongly disagree / Disagree / Agree / Strongly agree.
  The more participants agree or completely agree, the better the outcome

CONTACTS AND LOCATIONS:
Overall Officials: Michelle White, MD/MPH, Principal Investigator — Duke Health
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
If we plan to share with other researchers in the future, we will submit an amendment to the IRB.